CLINICAL TRIAL: NCT03235297
Title: Effects of Altitude on Single-Breath Diffusing Capacity for Carbon Monoxide in Normal Subjects and Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Altitude on Single-Breath Diffusing Capacity for Carbon Monoxide
Acronym: DLCO
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Matthew Hegewald, Adjunct Associate Professor, University of Utah, Intermountain Health Care, Inc.
Other Study IDs: DLCO
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: COPD
Keywords: Altitude; Diffusing capacity for carbon monoxide; COPD; Pulmonary function testing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Healthy subjects
- Subjects with COPD: Subjects with a diagnosis of COPD

SUMMARY:
The purpose of this study is to further understand the effects of altitude on the physiology of gas exchange in the pulmonary microcirculation in normal subjects and in people with chronic obstructive pulmonary disease (COPD) measured as the single-breath diffusing capacity for carbon monoxide (DLCOsb). The study will determine a mathematical formula to allow for altitude corrections in both study populations to be used clinically in pulmonary labs.

DETAILED DESCRIPTION:
The DLCOsb is one of the most common and widely tests clinically used across the world in pulmonary function laboratories to assess gas exchange from the lung to hemoglobin in the pulmonary circulation. This test is used in the differential diagnosis of respiratory related symptoms, to grade the degree of severity in lung disease, and to objectively monitor the progression of disease or the response to therapies. Therefore, it is important to have standard methods of performing and interpreting this test.This is a prospective study, collecting data from subjects at different simulated altitudes. The study hypothesis is that increasing altitude will increase the DLCOsb in a predictable manner that will allow for mathematical corrections to be applied for uniform interpretation in pulmonary labs at differing altitudes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20- 80 years
* Subjects must be either healthy or have been diagnosed with COPD

Exclusion Criteria:

* Anemia (hemoglobin < 10.0 g/dL)
* Carboxyhemoglobin > 3%
* Active smoking
* Heart disease or heart failure
* Pulmonary hypertension
* COPD exacerbation
* Pneumothroax within 6 months
* Bullous emphysema on chest imaging (Chest X-ray or CT)
* Supplemental oxygen use
* Diabetes mellitus
* Alcohol dependence
* Non-English speaking

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women, ages 20-80, both healthy subjects and those with a diagnosis of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Effect of altitude on measured diffusing capacity for carbon monoxide | 3 weeks

SECONDARY OUTCOMES:
Comparison of a novel inert gas technique for measuring alveolar volume with body plethysmography | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hegewald, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hegewald MJ, DeCato TW, Weaver LK, Jensen RL. Effect of barometric pressure on single-breath carbon monoxide diffusing capacity. Respir Physiol Neurobiol. 2023 Feb;308:103997. doi: 10.1016/j.resp.2022.103997. Epub 2022 Nov 17. PMID 36402362